CLINICAL TRIAL: NCT03091101
Title: Impact of Scleral Contact Lens Wear on Corneal Sensitivity, Nerve Morphology and Inflammation in Keratoconic Eyes
Brief Title: Impact of Scleral Contact Lens Wear on Corneal Nerves in Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Precision Technology Services Ltd (Unknown)
Responsible Party: Principal Investigator, Edward Lum, Post-Doctorial Fellow, University of Waterloo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ORE#21910
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Keratoconus
Keywords: keratoconus; corneal innervation; scleral contact lenses
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Scleral lens wearing keratoconics (Experimental): Newly diagnosed keratoconics with no previous rigid lens wear fitted with Sceral contact lenses
  Interventions: Device: Scleral lens wearing keratoconics

INTERVENTIONS:
Device: Scleral lens wearing keratoconics — Cohort of keratoconics fitted with scleral lenses and monitored over 6 months

SUMMARY:
The purpose of this study is to investigate changes in corneal innervation during scleral contact lens wear in a keratoconic population. Specifically, changes in corneal sensitivity and nerve fiber density from baseline in the central and mid-peripheral corneal locations will be measured over a 6-month lens wear period. An additional aim of the study is to investigate the impact of scleral lens wear on corneal inflammation within the same study group. This will be achieved by comparing dendritic cell density change from baseline over the study period.

DETAILED DESCRIPTION:
The human cornea is a densely innervated tissue that provides a high level of sensitivity to foreign objects or noxious substances. The innervation of the cornea also plays an important role in the tropic maintenance and repair of the corneal surface. Any alterations to the normal innervation of the cornea not only lessen the ability to detect foreign objects that could damage the ocular surface, but also reduce its wound healing ability. Previous studies have shown rigid contact lens wear reduces corneal sensitivity and nerve fiber density in keratoconic subjects. Scleral contact lenses are large diameter rigid gas permeable lenses that rests on the sclera while vaulting over the cornea with a fluid reservoir. The use of scleral contact lenses is becoming one of the current standard nonsurgical management of corneal dystrophies such as keratoconus, mainly due to the improved comfort and vision quality compared to conventional rigid lenses. Despite these patient benefits, little is known about the impact of scleral contact lens wear on corneal sensitivity and nerve morphology in keratoconus.

The purpose of this study is to investigate changes in corneal innervation during scleral contact lens wear in a keratoconic population. Specifically, changes in corneal sensitivity and nerve fiber density from baseline in the central and mid-peripheral corneal locations will be measured over a 6-month lens wear period. An additional aim of the study is to investigate the impact of scleral lens wear on corneal inflammation within the same study group. This will be achieved by comparing dendritic cell density change from baseline over the study period.

The investigators propose to take a sample of keratoconic participants and fit them in scleral lenses and:

1. Measure corneal sensitivity at two corneal locations before and after 1-month, 3-months and 6-months of scleral lens wear.
2. Capture images of the sub-basal nerve plexus in vivo using laser-scanning confocal microscopy at similar corneal locations and study visits.
3. Calculate nerve morphology parameters and dendritic cell density from these captured images.

Up to 15 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Had been diagnosed with keratoconus in at least one eye.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.

Exclusion Criteria:

* Have worn rigid corneal lenses for more than several days over the past year
* Is using any topical medications that will affect ocular health.
* Has any ocular pathology or systemic disease that may lead to severe insufficiency of lacrimal secretion (severe dry eyes) or corneal hypoesthesia which would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities and active neovascularization.
* Is aphakic.
* Has undergone any corneal surgery.
* Is participating in any other type of eye related clinical or research study.
* Has any known allergies or sensitivity to the diagnostic pharmaceuticals or products, such as fluorescein and topical anesthetics, used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Corneal sensitivity | 6-month lens wear period
  Indication of functional change in corneal innervation from scleral lens wear by measuring change in sensitivity threshold (grams/sq.mm) over time
Subbasal nerve fiber density | 6-month lens wear period
  Indication of morphological change in corneal innervation from scleral lens wear by measuring nerve fiber density changes (mm/sq.mm) in the central subbasal nerve fiber layer location over time.

SECONDARY OUTCOMES:
Corneal inflammation | 6-month lens wear period
  Changes in dendritic cell density (number/sq.mm) as a marker of corneal inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lum, PhD, Principal Investigator — Univerity of Waterloo
Locations (1):
- School of Optometry and Vision Science, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided